CLINICAL TRIAL: NCT07403357
Title: Effects of Stomatognathic Alignment Exercise Program in Craniomandibular Dysfunction.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0186
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Craniomandibular Dysfunction
Keywords: functional disability; Temporomandibular joint; Forward head posture; Myofascial release; Stomatognathic Alignment Exercise; Stomatognathic disease; Craniomandibular Dysfunction
MeSH Terms: conditions — Stomatognathic Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stomatognathic alignment exercise program along with standard physical therapy (Experimental): Stomatognathic alignment exercise program along with standard treatment.
  Interventions: Other: Stomatognathic Alignment Exercise Program; Other: Standard Physical therapy treatment
- Traditional physical therapy (Active Comparator): Myofascial release of masticatory muscles and heating pad at cervical.
  Interventions: Other: Standard Physical therapy treatment

INTERVENTIONS:
Other: Stomatognathic Alignment Exercise Program — Chin Tuck Exercise:
  Starting position: Supine and standing against a wall. Tuck chin backward over the sternal notch to place the patient's ears in line with the tips of the shoulders.
  Repetitions:
  Supine: Ten repetitions of a 10-second hold. Standing against a wall: Two repetitions of a 5-minute hold.
  Anterior Chest Stretching Exercise:
  Starting position: Standing against a wall with a flattened back; arms at 45° shoulder abduction with elbow in full extension.
  Active ROM exercises of neck and TMJ:
  Starting position: Sitting in a back-supported chair. Neck motions: flexion, extension, lateral flexion, and rotation. TMJ: Mouth opening, lateral excursion, and protrusion. Repetitions: A 10-second hold at the end range of each motion. Two series of ten repetitions for each motion.
  Standard physiotherapy including hot pack and myofascial release of masticatory muscles.
  A total of 12 sessions were conducted for 4 weeks with 3 sessions scheduled each week.
  Arms: Stomatognathic alignment exercise program along with standard physical therapy
Other: Standard Physical therapy treatment — Control Group received only standard physiotherapy including hot pack and myofascial release of masticatory muscles. A total of 12 sessions were conducted for 4 weeks with 3 sessions scheduled each week.

SUMMARY:
The study was conducted to determine the effects of stomatognathic alignment exercise program in craniomandibular dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Male and female with age group of 20-65 years.
* Patients diagnosed with temporomandibular dysfunction
* Individuals with the sedentary life style
* Craniovertebral angle <50 degrees
* Patients who presented with at least one symptom of temporomandibular dysfunction, able to communicate effectively, cooperative with imaging examinations, and able to complete the prescribed treatment and patients with no contraindications for the required examinations or treatments.

Exclusion Criteria:

* Serious musculoskeletal problems of cervical and thoracic spine
* Neurological disease affecting balance and postural control
* Dental prosthesis
* Disc prolapsed
* Previous surgery in TMJ area
* Vertebral artery compromise test
* Cerebrovascular disease

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | From enrollment until the end of treatment at the fourth week.
  Numeric Pain Rating Scale is utilized to evaluate pain. It consists of 11 points, having an overall score ranging from 0 to 10, where; 0 represents no pain, 1 to 3 represents mild pain, 4 to 6 represents moderate pain and 7 to 10 represents the most severe pain.
Mandibular function impairment questionnaire | From enrollment until the end of treatment at the fourth week.
  MFIQ is used to evaluate the degree of jaw function impairment in TMJD patients. Two dimensions and 17 questions make up this questionnaire, which assigns a score ranging from 0 (no problem) to 4 (extreme difficulty or impossible without support) for a certain jaw function. The "functional capacity" dimension is made up of the first eleven components, whereas the "nutrition" dimension is made up of the next six. A high degree of jaw function impairment is indicated by a high overall score on the questionnaire.

SECONDARY OUTCOMES:
ROM Cervical Spine (Felxion) | From enrollment until the end of treatment at the fourth week
  Changes in cervical spine flexion ROM at baseline and 4th week of intervention was measured using goniometer.
ROM Cervical Spine (Extension) | From enrollment until the end of treatment at the fourth week.
  Changes in cervical spine extension ROM at baseline and 4th week of intervention was measured using goniometer.
ROM Cervical Spine (Lateral Flexion) Left Side | From enrollment until the end of treatment at the fourth week.
  Changes in cervical spine lateral flexion on left side ROM at baseline and 4th week of intervention was measured using goniometer.
ROM Cervical Spine (Lateral Flexion) Right Side | From enrollment until the end of treatment at the fourth week.
  Changes in cervical spine lateral flexion on right side ROM at baseline and 4th week of intervention was measured using goniometer.
ROM Cervical Spine (Rotation) Left Side | From enrollment until the end of treatment at the fourth week.
  Changes in cervical spine rotation on left side ROM at baseline and 4th week of intervention was measured using goniometer.
ROM Cervical Spine (Rotation) Right Side | From enrollment until the end of treatment at the fourth week.
  Changes in cervical spine rotation on right side ROM at baseline and 4th week of intervention was measured using goniometer.
ROM temporomandibular joint, mouth opening (Depression) | From enrollment until the end of treatment at the fourth week.
  Changes in mouth opening ROM at baseline and 4th week of intervention was measured using ruler.
ROM temporomandibular joint (Protrusion) | From enrollment until the end of treatment at the fourth week.
  Changes in protrusion ROM at baseline and 4th week of intervention was measured using ruler.
ROM temporomandibular joint (Lateral Excursion) Left side | From enrollment until the end of treatment at the fourth week.
  Changes in lateral excursion on left side ROM at baseline and 4th week of intervention was measured using ruler.
ROM temporomandibular joint (Lateral Excursion) Right side | From enrollment until the end of treatment at the fourth week.
  Changes in lateral excursion on right side ROM at baseline and 4th week of intervention was measured using ruler
Craniovertebral angle | From enrollment until the end of treatment at the fourth week.
  For assessing the severity and alignment of forward head posture by evaluating the position of the head in relation to the trunk. Changes in craniovertebral angle at baseline and 4th week of intervention was measured using Markus Bader-Software solution.

CONTACTS AND LOCATIONS:
Overall Officials: Saba Rafique, MS.OMPT, Principal Investigator — Riphah International University
Locations (1):
- Fatima Memorial Hospital (Oral & Maxillofacial Surgery Department), Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oh DW, Kang TW, Kim SJ. Effect of stomatognathic alignment exercise on temporomandibular joint function and swallowing function of stroke patients with limited mouth opening. J Phys Ther Sci. 2013;25(10):1325-9
- [Background] Pundkar S, Patil D, Naqvi W. A Comparative Study on Effectiveness of Rocabado Approach and Conventional Physiotherapy on Pain, ROM and QOL in Patients with TMJ Dysfunction. Journal of Pharmaceutical Research International. 2021;33(58B):201-9
- [Background] Byra J, Kulesa-Mrowiecka M, Pihut M. Physiotherapy in hypomobility of temporomandibular joints. Folia Med Cracov. 2020;60(2):123-34
- [Background] Oleksy Ł, Kielnar R, Mika A, Jankowicz-Szymańska A, Bylina D, Sołtan J, et al. Impact of Cervical Spine Rehabilitation on Temporomandibular Joint Functioning in Patients with Idiopathic Neck Pain. Biomed Res Int. 2021;2021:6886373
- [Background] Yılmaz V, Aras B, Umay E. Temporomandibular Joint Dysfunction and Impaired Stomatognathic Alignment: A Problem Beyond Swallowing in Patients With Stroke. Indian J Otolaryngol Head Neck Surg. 2020;72(3):329-34
- [Background] Militi A, Bonanno M, Calabrò RS. It Is Time for a Multidisciplinary Rehabilitation Approach: A Scoping Review on Stomatognathic Diseases in Neurological Disorders. J Clin Med. 2023;12(10)
- [Background] de Oliveira-Souza AIS, do Valle Sales LR, de Fontes Coutinho AD, de Oliveira DA, Armijo-Olivo S. Effectiveness of an 8-week neck exercise training on pain, jaw function, and oral health-related quality of life in women with chronic temporomandibular disorders: a randomized controlled trial. J Oral Facial Pain Headache. 2024;38(1):40-51
- [Background] Ilhanlı M, Ilhanlı I, Aksakallı S. Effectiveness of Rocabado exercises in patients with rheumatoid arthritis in remission with temporomandibular joint involvement: A randomized-controlled study. Turk J Phys Med Rehabil. 2024;70(3):319-26
- [Background] O. W. Conservative Management of Temporomandibular Joint Dysfunction: A Case Report. Journal of Health Directories. 2024;1(1):16-23
- [Background] Yu LJ, Yan X, Kim TH. Effects of combined jaw and cervicoscapular exercises on mouth opening and muscle properties in cervical extension type. Sci Rep. 2025;15(1):19049.